CLINICAL TRIAL: NCT03227679
Title: Metabolism-informed Care for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Hilary Tindle, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 160512
Record Dates: First submitted 2017-06-29; First posted 2017-07-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Use; Tobacco Use Cessation
Keywords: Personalized Medicine; Nicotine Metabolite Ratio (NMR); Varenicline; Nicotine Replacement Therapy (NRT); Smoking Cessation; Pharmacotherapy
MeSH Terms: conditions — Tobacco Use; Tobacco Use Cessation; Smoking Cessation | interventions — Varenicline; Bupropion; Tobacco Use Cessation Devices; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: Parallel arm pilot trial with a single-arm crossover design
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant, Nurse, and RAs all blinded to random Arm assignment, none blinded to medication prescription
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metabolism-Informed Care (MIC) (Active Comparator): Smoking Cessation Pharmacotherapy (varenicline, bupropion, and nicotine patch) recommendations were guided by Nicotine Metabolism as measured by the Nicotine Metabolite Ratio. Ultimately, after being educated about smoking cessation medication efficacy and side-effects, the participant could decide to take any medication for which they were medically cleared, but the recommendation was made based on rate of Nicotine Metabolism.
  Interventions: Other: Nicotine Metabolite Ratio; Drug: Varenicline; Drug: Bupropion; Drug: Nicotine patch
- Guideline-Based Care (GBC) (Active Comparator): Smoking Cessation Pharmacotherapy (varenicline, bupropion, and nicotine patch) was co-selected from those they were medically able to receive after educating participants about smoking cessation medication efficacy and side-effects.
  Interventions: Drug: Varenicline; Drug: Bupropion; Drug: Nicotine patch

INTERVENTIONS:
Other: Nicotine Metabolite Ratio — This intervention used information from a genetically-informed biomarker (Nicotine Metabolite Ratio, NMR) to assign one of 3 FDA-approved smoking cessation pharmacotherapies (varenicline, bupropion, or NRT) to participants.
  Arms: Metabolism-Informed Care (MIC)
Drug: Varenicline — FDA-approved smoking cessation pharmacotherapy
  Other Names: Chantix
Drug: Bupropion — FDA-approved smoking cessation pharmacotherapy
  Other Names: Zyban
Drug: Nicotine patch — FDA-approved smoking cessation pharmacotherapy
  Other Names: Nicotine Replacement Therapy (NRT)

SUMMARY:
Nicotine mediates smoking's addictive effects in the brain. The ratio of 3-hydroxycotinine to cotinine, known as the nicotine metabolite ratio, or NMR, is a genetically- informed biomarker reflecting hepatic CYP2A6 activity and the rate of nicotine metabolism. In light of a recent randomized controlled trial (RCT) in humans in Lancet Respiratory Medicine, which found that the NMR can be used to individualize treatment for smokers, our pilot study aims to determine the feasibility of using NMR to guide selection of pharmacotherapy in clinical populations of daily smokers.

DETAILED DESCRIPTION:
Consenting participants will be assigned to guideline-based care (GBC: incorporating national guidelines and more recent evidence from clinical trials of pharmacotherapy for smoking cessation) or metabolism-informed care (MIC: identical to GBC but selection of medication based on NMR result). All participants received counseling from a nurse level certified tobacco counseling. After consent, participants undergo a blood draw for NMR, complete a baseline questionnaire, and are randomized to GBC or MIC. At approximately 1, 3, and 6 months post-consent, participants will provide follow up information via telephone questionnaire regarding symptoms, confidence in quitting, use of medications, and smoking status. At the 6-month follow-up time point, if a participant self-reports abstinence from smoking, the participant will be asked to complete a survey in-person and provide a sample of end-expired carbon monoxide for biochemical validation. At the 6 month time point, GBC participants who continue to smoke will be offered an additional phone call from the nurse tobacco counselor in which the results of the baseline NMR test will be given, along with a second prescription for a smoking cessation medication based on the NMR results (i.e., single arm crossover design). Two weeks after this additional phone call, the patient will be contacted for a final survey regarding use of medication and smoking status.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Smokes ≥ 5 cigarettes per day
* Willing to give up all forms of tobacco (5/10/2016 - 6/27/2016)
* Medically cleared (i.e., no contraindications in Section 3) to receive at least 2 FDA- approved smoking cessation medications
* Willing to use the medications for which medically cleared (individually, not in combination; only applicable if Medically Cleared = Yes)

Exclusion Criteria:

* Current diagnosis of schizophrenia, psychosis, active suicidal ideation, dementia, or severe mental retardation
* Receiving palliative or hospice care
* Currently pregnant or breastfeeding
* Hospitalized for a psychiatric condition in the past year (5/10/2016 - 6/27/2016)
* Hospitalized for a psychiatric condition in the past 3 months or change in psychiatric medications in last 3 months (6/28/2016 forward)
* Telephone problems that would preclude participation (e.g., can't receive calls reliably)
* Not able to read and speak English
* Abstinent from cigarettes for >3 days (b/c NMR not reliable after 72 hours)
* Used smoking cessation medications in the last 7 days (5/10/2016 - 6/27/2016)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2016-10-08 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Theoretical Endorsement of MIC as assessed by level of agreement to a set of seven 5-point Likert Scale questions | Baseline
  Likert Scale from Strongly Disagree to Strongly Agree on items assessing attitudes toward and perceptions of using metabolism information to guide medical care
Acceptance of MIC medication recommendation as assessed by concordance between MIC recommendation and actual prescribed medication | At 4 weeks post-baseline
  Level of agreement between participant's prescribed medication and the medication that would be recommended based on Nicotine Metabolite Ratio

SECONDARY OUTCOMES:
Confidence in Quitting | Baseline - 6 months
  Self-reported confidence in ability to quit
Medication Use/Compliance | 1 - 6 months
  Use of prescribed medication, as directed
Smoking Status | 6 months
  Self-reported and/or biochemically validated smoking cessation

CONTACTS AND LOCATIONS:
Overall Officials: Quinn Wells, MD, Principal Investigator — Vanderbilt University Medical Center; Dawn Beaulieu, MD, Principal Investigator — Vanderbilt University Medical Center; Matthew Freiberg, MD, Principal Investigator — Vanderbilt University Medical Center; Hilary Tindle, MD, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. Assessment of the Economic Costs of Smoking. Economics of tobacco toolkit. 2011;:1-116.
- [Background] Agaku IT, King BA, Dube SR; Centers for Disease Control and Prevention (CDC). Current cigarette smoking among adults - United States, 2005-2012. MMWR Morb Mortal Wkly Rep. 2014 Jan 17;63(2):29-34. PMID 24430098
- [Background] Benowitz NL. Pharmacology of nicotine: addiction, smoking-induced disease, and therapeutics. Annu Rev Pharmacol Toxicol. 2009;49:57-71. doi: 10.1146/annurev.pharmtox.48.113006.094742. PMID 18834313
- [Background] Hukkanen J, Jacob P 3rd, Benowitz NL. Metabolism and disposition kinetics of nicotine. Pharmacol Rev. 2005 Mar;57(1):79-115. doi: 10.1124/pr.57.1.3. PMID 15734728
- [Background] Chen LS, Bloom AJ, Baker TB, Smith SS, Piper ME, Martinez M, Saccone N, Hatsukami D, Goate A, Bierut L. Pharmacotherapy effects on smoking cessation vary with nicotine metabolism gene (CYP2A6). Addiction. 2014 Jan;109(1):128-137. doi: 10.1111/add.12353. Epub 2013 Nov 11. PMID 24033696
- [Background] Dempsey D, Tutka P, Jacob P 3rd, Allen F, Schoedel K, Tyndale RF, Benowitz NL. Nicotine metabolite ratio as an index of cytochrome P450 2A6 metabolic activity. Clin Pharmacol Ther. 2004 Jul;76(1):64-72. doi: 10.1016/j.clpt.2004.02.011. PMID 15229465
- [Background] Lerman C, Schnoll RA, Hawk LW Jr, Cinciripini P, George TP, Wileyto EP, Swan GE, Benowitz NL, Heitjan DF, Tyndale RF; PGRN-PNAT Research Group. Use of the nicotine metabolite ratio as a genetically informed biomarker of response to nicotine patch or varenicline for smoking cessation: a randomised, double-blind placebo-controlled trial. Lancet Respir Med. 2015 Feb;3(2):131-138. doi: 10.1016/S2213-2600(14)70294-2. Epub 2015 Jan 12. PMID 25588294
- [Background] Hughes JR, Stead LF, Hartmann-Boyce J, Cahill K, Lancaster T. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2014 Jan 8;2014(1):CD000031. doi: 10.1002/14651858.CD000031.pub4. PMID 24402784
- [Background] Bauld L, Bell K, McCullough L, Richardson L, Greaves L. The effectiveness of NHS smoking cessation services: a systematic review. J Public Health (Oxf). 2010 Mar;32(1):71-82. doi: 10.1093/pubmed/fdp074. Epub 2009 Jul 28. PMID 19638397
- [Background] 2008 PHS Guideline Update Panel, Liaisons, and Staff. Treating tobacco use and dependence: 2008 update U.S. Public Health Service Clinical Practice Guideline executive summary. Respir Care. 2008 Sep;53(9):1217-22. No abstract available. PMID 18807274
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Anthenelli RM, Benowitz NL, West R, St Aubin L, McRae T, Lawrence D, Ascher J, Russ C, Krishen A, Evins AE. Neuropsychiatric safety and efficacy of varenicline, bupropion, and nicotine patch in smokers with and without psychiatric disorders (EAGLES): a double-blind, randomised, placebo-controlled clinical trial. Lancet. 2016 Jun 18;387(10037):2507-20. doi: 10.1016/S0140-6736(16)30272-0. Epub 2016 Apr 22. PMID 27116918

DOCUMENTS (2):
  • Study Protocol (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT03227679/Prot_000.pdf
  • Informed Consent Form (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT03227679/ICF_001.pdf